CLINICAL TRIAL: NCT00966121
Title: RCT Comparing the Efficacies of Endoscopic Variceal Ligation (EBL) and Combined Treatment of Beta-blocker and EBL for the Prevention of Esophageal Variceal Rebleeding
Brief Title: Endoscopic Band Ligation (EBL) Versus Endoscopic Band Ligation and Propranolol for the Prevention of Variceal Rebleeding
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Soon Ho Um, Professor, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EBLPPL-1
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Cirrhosis; Variceal Bleeding
Keywords: Cirrhosis; Esophagus Disorders; Varicose Veins
MeSH Terms: conditions — Fibrosis; Esophageal Diseases; Varicose Veins

STUDY DESIGN:
Intervention Model Description: Endoscopic Band Ligation (EBL) Versus Endoscopic Band Ligation and Propranolol
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic band ligation (Active Comparator): Perform endoscopic band ligation (EBL) until esophageal varices are eradicated, and then follow-up endoscopy with 3-6 months interval
  Interventions: Procedure: endoscopic band ligation
- EBL+Propranolol (Active Comparator): Perform EBL same as EBL group. In addition, take propranolol to reduce 25% in HR or HR ≤55/min
  Interventions: Procedure: EBL+Propranolol

INTERVENTIONS:
Procedure: endoscopic band ligation — * Perform EBL within 7 days after randomization
  * Apply 1-2 band/column/session to varices in the distal 5-7cm of the esophagus till they are eradicated (Disappearance or too small to apply band) with interval of 4weeks (at 4,8,12 weeks after initial treatment).
  * Acid suppression using proton pump inhibitor until eradicated.
  * After eradication, then follow-up endoscopy according to a preset schedule (at 1, 2, 3 months after initial treatment, then every 3-6 months until 36 months).
  Arms: Endoscopic band ligation
Procedure: EBL+Propranolol — * Start with 20 mg b.i.d
  * Adjust by 20-40 mg/d reaching reduction by 25% in HR or HR ≤55/min
  * After reaching target HR, then FU according to a preset schedule (at 1, 2, 3 months after initial treatment, then every 3 months until 36 months)
  Arms: EBL+Propranolol

SUMMARY:
Both propranolol and endoscopic band ligation (EBL) are effective for prevention of variceal rebleeding. Recently several studies compared the efficacy of EBL alone and with a combination of propranolol and EBL. However, the results of recent studies showed discrepancy. This study is performed to compare the efficacy and safety of EBL alone and EBL combined with propranolol in patients without previous history of endoscopic variceal treatment.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* age between 18 and 70 years
* Successful control of esophageal variceal bleeding within 6 weeks before enrollment

Exclusion Criteria:

* Gastric variceal bleeding
* Patients with systolic blood pressure <100 mmHg or basal heart rate <60/min
* Portal vein thrombosis
* Prominent hepatic encephalopathy
* Coexisting untreated malignancy
* Severe cerebrovascular or cardiovascular disease, renal failure
* Previous history of endoscopic, radiologic, or surgical treatment for varices or ascites
* Contraindication to beta-blocker
* Pregnancy
* Refusal to give consent to participate in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2008-08; Primary Completion 2019-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Rebleeding from esophageal varices | 2 years
  Rebleeding from esophageal varices

SECONDARY OUTCOMES:
Upper gastrointestinal bleeding; significant esophageal variceal bleeding; mortality;adverse events | 2 years
  Upper gastrointestinal bleeding; significant esophageal variceal bleeding; mortality;adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea